CLINICAL TRIAL: NCT05774834
Title: A Non-interventional Functional Magnetic Resonance Imaging (fMRI) Study on the Neural Bases of Decision-making in Healthy Individuals
Brief Title: Neural Bases of Decision-making in Healthy Individuals
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 2137
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: decision-making; executive functioning; fMRI; ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All healthy participants: All healthy participants will undergo behavioral assessment and fMRI
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this single center non-interventional fMRI study is to assess the neural bases of decision-making and executive functioning in healthy individuals,and whether/how their responsiveness is modulated by ageing. The main questions it aims to answer are:

1. are there specific neural correlates for ageing effects on executive functioning (particularly inhibitory control) and decision-making?
2. Is there a relationship, at the behavioral and neural levels, between ageing-related changes in executive functioning and decision-making?

Healthy participants will be recruited for

1. a behavioral assessment including multiple tests of decision-making and executive functioning/inhibitory control;
2. a fMRI session to collect data concerning a) brain activity associated with decision-making and executive functioning, b) brain structural morphometriy (grey-matter volume/density), and c) brain structural connectivity (diffusion weighted imaging).

Results will provide an useful baseline for investigating alterations of decision-making and executive functioning, and of their neural bases, in pathological conditions.

DETAILED DESCRIPTION:
The fast growth of Decision Neuroscience is contributing to unveil the cognitive processes underlying choices and their neural bases. The results obtained so far show that decision-making involves neural mechanisms underpinning a complex balance between automatic appetitive or aversive drives generated by subcortical structures, and processes of executive control centered in fronto-parietal brain networks. While the role of meso-limbic structures in reinforcement learning have been widely investigated, it is much less clear to what extent are choices shaped by a) individual differences in executive skills; b) contextual factors potentially interfering with such skills, such as knowing that the outcome of those choices will impact only on one's own vs. another's welfare. This a critical gap, since executive abilities are known to decline even in physiological ageing, thus potentially interfering with the quality of choices. On this ground, this single center non-interventional fMRI study aims to provide novel insights into the relationship between executive and decision-making skills, and their possible changes with ageing, in 150 healthy individuals. This goal will be pursued by combining a behavioral assessment of decision-making and executive skills with a multimodal fMRI session including data concerning a) brain activity associated with decision-making and executive functioning in social vs. non-social contexts, b) brain structural morphometry (grey-matter volume/density), and c) brain structural connectivity (diffusion weighted imaging). The behavioral assessment will involve the main metric of decision-making (e.g., risk aversion, loss aversion, delay discounting) and executive functioning (e.g., selective attention and inhibitory control). MRI data will unveil the neural bases of individual differences in decision-making and executive performance in terms of performance-related patterns of brain activity, structure and connectivity. Results will provide an useful baseline for investigating alterations of decision-making and executive functioning, and of their neural bases, in pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, as determined by screening assessments and principal investigator judgment
* The participant must be able to comply with study requirements as judged by the principal investigator

Exclusion Criteria:

* Any history of alcohol and/or drug abuse, addiction or suspicion of regular consumption of drugs of abuse
* Use of any psychoactive medication, or medications known to have effect on central nervous system (CNS) or blood flow
* Any contraindications for magnetic resonance imaging (MRI) scans or any brain/head abnormalities restricting MRI eligibility

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 150 healty individuals, aged 18-60 years, sampled from the general population
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral performance 1: Decision-making skills | MRI-acquisition day 1
  Participants' decision-making performance will be assessed in terms of "loss aversion" (i.e., the overweighting of potential losses compared with gains), after removing the potential confounding effect of risk aversion

SECONDARY OUTCOMES:
Behavioral performance 2: Executive functioning skills | MRI-acquisition day 1
  Participants' executive performance will be assessed in terms of well-know metrics such as selective attention and inhibitory control, measured with the Stroop Task and the Stop-Signal-Task, respectively.
Brain activity underlying decision-making and executive performance | MRI-acquisition day 1
  Standard pipelines and pre-processing of fMRI task-related data will be used to detect regional changes of brain activity associated with individual differences in decision-making and executive performance.
Brain structure related to decision-making and executive performance | MRI-acquisition day 1
  Standard pipelines and pre-processing of MRI T1-weighted data will be used to detect patterns of GM volume/density and structural connectivity associated with individual differences in decision-making and executive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Ita, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing will assessed case by case, and data will be made available on reasonable request.